CLINICAL TRIAL: NCT05549479
Title: A Pilot Randomized Controlled Trial of a Virtual Peer-support Exercise Intervention for Older Adults with Cancer
Brief Title: Virtual Peer-support Exercise Intervention for Older Adults with Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: JST-3
Record Dates: First submitted 2022-08-23; First posted 2022-09-22 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-01

CONDITIONS: Cancer; Aging
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (AgeMatchPLUS). (Experimental)
  Interventions: Behavioral: Peer Matching; Behavioral: Qualified Exercise Professional Support Sessions
- Control Condition (AgeMatch): (Active Comparator)
  Interventions: Behavioral: Peer Matching

INTERVENTIONS:
Behavioral: Peer Matching — Participants will be matched with a peer based on evidence informed criteria. Partners will independently communicate and support each other around exercise for the duration of the study.
Behavioral: Qualified Exercise Professional Support Sessions — Dyads will participate in weekly virtual sessions with a QEP for 10 weeks. Each session will last up to 1 hour. The QEP (i.e., registered kinesiologist) will provide a tailored exercise program, focusing on aerobic activity for both individuals in the dyad based on personal circumstances, cancer-related characteristics, side effects, current fitness level (consistent with home-based exercise strategies), and personal preferences.
  Arms: Intervention Group (AgeMatchPLUS).

SUMMARY:
Background:

By 2030, 23% of Canadians will be over 65 years of age. Two in five of these individuals will be diagnosed with cancer. Older adults have high levels of functional decline, and a cancer diagnosis adds prolonged physical sequelae to the natural aging process. Many of these effects can be mitigated by regular exercise. However, older adult cancer survivors are significantly less likely to meet current exercise guidelines than their younger counterparts. As our population ages, we need to develop effective, scalable interventions that support health in older adult cancer survivors. The objective of this study is to determine the feasibility and preliminary effectiveness of a virtually delivered peer exercise intervention with qualified exercise professional (QEP) support for older adult cancer survivors.

Methods:

Participants will include older adult cancer survivors who are cleared for exercise, have consistent access to the internet, and currently take part in less than 150 minutes of exercise per week. All participants will be matched with a partner, given a peer support guide, and information on current exercise guidelines. In addition to being matched with a peer, dyads in the intervention group will have weekly virtual sessions with a QEP for 10 weeks. Participants in the control group will independently support their partner around exercise for 10 weeks.

Outcomes:

Participants will be assessed at 3 time points. The primary outcome is feasibility. This will be measured by assessing recruitment, retention, adherence rates to the intervention, and participant acceptability and satisfaction. Secondary effectiveness outcomes include exercise volume, social support, quality of life, physical function, and physical activity enjoyment.

Impact:

If effective, this will be the first virtual peer-based exercise intervention for older adult cancer survivors. Findings will inform future methods aimed at increasing exercise in older adults.

DETAILED DESCRIPTION:
METHODS

Research Questions:

Research Question 1 (primary). Is a virtually-delivered, peer matching exercise intervention supported by qualified exercise professionals (QEP) feasible for older adult cancer survivors? Research Question 2. Do older adult cancer survivors who participate in a virtually-delivered peer matching exercise intervention with QEP support have improved levels of social support compared to those matched with a peer only? Research Question 3. Do older adult cancer survivors who participate in a virtually-delivered peer matching exercise intervention with QEP support have improved levels of physical activity behaviour, health-related quality of life and physical functioning compared to those who are matched with a peer only?

Study Design:

This is a two-arm pilot randomized controlled trial with blinded outcome assessment. The protocol and study methods adhere to the CONSORT extension for randomized pilot trials. The Hamilton Integrated Research Ethics Board will approve this study. Dyads will be randomized (1:1) to the Intervention (AgeMatchPLUS) or control (AgeMatch) groups prior to baseline assessment. Group allocation will be centrally randomized using a web platform (https://www.randomizer.org/) by a graduate student external to the research team. A Research Assistant will assign group allocation in the order participants complete an initial demographics questionnaire and are matched with a peer for the study.

Intervention:

Peer Matching. A Research Assistant will match all participants into dyads based on evidence-informed criteria. To be matched, females must be in the same time zone and diagnosed with the same type of cancer. Matched peers will be introduced to each other by a Research Assistant via zoom after baseline data collection. All participants will be given a peer support guide that provides tips for supporting their exercise partner, an infographic on exercise guidelines for older cancer survivors and a Fitbit Inspire 2©. Partners will independently communicate and support each other around exercise for the duration of the study.

Intervention Group (AgeMatchPLUS). This group will have dyads participate in weekly virtual sessions with a QEP for 10 weeks. Each session will last up to 1 hour. The QEP (i.e., registered kinesiologist) will provide a tailored exercise program, focusing on aerobic activity with both participants in the dyad based on personal circumstances, cancer-related characteristics, side effects, current fitness level, and personal preferences. Overall, content discussed at the sessions will include a review of the exercise program, barriers to exercise participation, achievement of goals, and adverse events. For four weeks following the 10-week intervention, the QEP will be available for consultation (labelled "tapering" period) as needed by participants in this group. This tapering period is important to understand strategies to successfully taper older adults from an exercise trial. Also, during the tapering period, participants in this group will receive two supportive emails from the QEP encouraging ongoing maintenance of exercise and social support.

Control Condition (AgeMatch): Dyads in this group will independently communicate and support each other around exercise for 10 weeks. They will not have contact with the QEP during the intervention or tapering period and will structure their communication (mode and frequency) with their matched peer.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Older adult (>60 years)
* Living with or beyond a cancer diagnosis (any type or stage of cancer at any stage of treatment)
* Living in Canada
* Medically cleared for exercise
* Have consistent access to an internet-connected device with webcam
* Currently take part in less than 150 minutes of MVPA per week

Exclusion Criteria:

* Self-report any contraindications to exercise
* Had recent (in the last 4 weeks) or have planned surgery of any kind (including reconstructive surgery) in the next 3 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 10 weeks
  The percentage of eligible individuals who expressed interest in the study that enrolled
Retention rate | 10 weeks
  The percentage of enrolled participants who completed the intervention
Adherence rate | 10 weeks
  The percentage of total sessions attended and tracked using weekly logs
Participant Satisfaction | 10 weeks
  7 points Likert satisfaction scale

SECONDARY OUTCOMES:
Exercise volume | 10 weeks
  Fitbit Inspire
Exercise volume | 14 weeks
  Fitbit Inspire
Exercise volume | 10 weeks
  Godin Leisure Time Exercise Questionnaire (higher scores represent higher volume of exercise)
Exercise volume | 14 weeks
  Godin Leisure Time Exercise Questionnaire (higher scores represent higher volume of exercise)
Social support | 10 weeks
  Social Support Survey (0-7 scale; higher scores indicate higher levels of social support)
Social support | 14 weeks
  Social Support Survey (0-7 scale; higher scores indicate higher levels of social support)
Health-related quality of life | 10 weeks
  Eq-5d-3L (5 dimensions each with a 3 level scale; lower scores indicate higher levels of quality of life)
Health-related quality of life | 14 weeks
  Eq-5d-3L (5 dimensions each with a 3 level scale; lower scores indicate higher levels of quality of life)
Self-report physical functioning | 10 weeks
  Patient Specific Functional Scale (10 point scale; higher scores represent higher quality of life)
Self-report physical functioning | 14 weeks
  Patient Specific Functional Scale (10 point scale; higher scores represent higher quality of life)
Sub-max aerobic capacity | 10 weeks
  Six minute walk test
Sub-max aerobic Capacity | 14 weeks
  Six minute walk test
Physical functioning | 10 weeks
  30 second sit to stand
Physical functioning | 14 weeks
  30 second sit to stand
Enjoyment of performing physical activity | 10 weeks
  Physical Activity Enjoyment Scale (7 point scale for each item; higher overall scores indicate higher enjoyment of physical activity)
Enjoyment of performing physical activity | 14 weeks
  Physical Activity Enjoyment Scale (7 point scale for each item; higher overall scores indicate higher enjoyment of physical activity)

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith-Turchyn J, Sinclair S, O'Loughlin EK, Innes A, Vani MF, Beauchamp M, Phillips SM, Richardson J, Thabane L, Sabiston CM. A pilot randomized controlled trial of a virtual peer-support exercise intervention for female older adults with cancer. BMC Geriatr. 2024 Oct 26;24(1):887. doi: 10.1186/s12877-024-05495-z. PMID 39462335